CLINICAL TRIAL: NCT04511143
Title: Investigation of the Correlation Between Ultrasonography Based Muscle Architecture Parameters and Maximum Voluntary Isometric Knee Flexor Muscle Strength
Brief Title: The Correlation Between Ultrasonography Based Muscle Architecture Parameters and Voluntary Isometric Muscle Strength
Status: Completed | Type: Observational
Sponsor: Istanbul Kültür University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Gülşah Karaca, Research Assistant, Istanbul Kültür University
Other Study IDs: Istanbul Kultur University
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Ultrasound Imaging
MeSH Terms: interventions — Muscle Strength

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: muscle strength and ultrasound imaging measurement — hamstring muscle strenght measured by hand held dynamometer. The long head of Biceps Femoris, Semitendinosus, Semimembronosus were evaluated by B-mode ultrasound imaging.

SUMMARY:
The goal of this study is to investigate potential relations of ultrasound-based muscle architecture parameters and isometric knee flexor muscle strength (IKFS) in healthy individuals. IKFS was measured for twenty participants (22.15±2.41 y.o; 8 females, 12 males) by a hand-held dynamometer. Investigated parameters were total and individual cross-sectional areas (CSA), Muscle-Thickness (MT), and pennation-angle (PA) for Biceps Femoris-long head (LBF), Semitendinosus (ST) and Semimembranosus (SM) muscles at 25%, 50% and 75% length of the thigh.

DETAILED DESCRIPTION:
The images of hamstring muscles were taken by a US device (Toshiba Aplio 500, Japan) with a linear probe (10-12 MHz, with a footprint of 52 mm).

For each participant, maximum voluntary IKFS was measured from the non-dominant side in the prone position with foot and ankle stayed outside of the bed. Maximum IKFS (20 limbs) was measured by an HHD (A Lafayette Model 01165) (Lafayette, IN) at 15° knee flexion in prone lying position

ELIGIBILITY:
Inclusion Criteria:

* being healthy young

Exclusion Criteria:

-

Ages: 20 Years to 28 Years | Sex: All
Age Groups: Adult
Study Population: Twenty healthy participants (22.15 ± 2.41 y.o; 1.72 ± 0.09 m; 66.5 ± 11.50 kg; 8 female, 12 male) participated in the study.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
The association between IKFS and ultrasound-based muscle architecture in this study will investigate potential relations of ultrasound-based muscle architecture parameters and isometric knee flexor muscle strength (IKFS) in healthy individuals. | an average of 1 year
  IKFS was measured for twenty participants by a hand-held dynamometer. Investigated parameters were total and individual cross-sectional areas (CSA), Muscle-Thickness (MT), and pennation-angle (PA) for Biceps Femoris-long head (LBF), Semitendinosus (ST) and Semimembranosus (SM) muscles at 25%, 50% and 75% length of the thigh. The association between IKFS and ultrasound-based muscle architecture parameters was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Nazıf E Akalan, Professor, Principal Investigator — Istanbul Kültür University; Bulent Bayraktar, Professor, Principal Investigator — Istanbul University; Sergen Devran, Researcher, Principal Investigator — Istanbul University; Omer B Gozubuyuk, M.D.,M.Sc.Dr, Principal Investigator — Istanbul University; Gulsah Karaca, Researcher, Principal Investigator — Istanbul Kültür University
Locations (1):
- Istanbul Kultur University, Istanbul, E5 Highway Bakırköy, İstanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided